CLINICAL TRIAL: NCT06422468
Title: Combining Accelerometer, Gyroscope, Sound, Electrocardiography and Photoplethysmography Data in Cardiac Monitoring: a Pilot Study
Brief Title: Combining Accelerometer, Gyroscope, Sound, Electrocardiography and Photoplethysmography Data in Cardiac Monitoring
Acronym: CARDS-pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z-2023103
Record Dates: First submitted 2024-02-08; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Photoplethysmography; Single-lead Electrocardiography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibriCheck recordings (Other)
  Interventions: Device: FibriCheck recordings

INTERVENTIONS:
Device: FibriCheck recordings — PPG, ACC, GYR, ECG and sound measurements

SUMMARY:
The goal of this interventional clinical trial is to investigate whether combining photoplethysmography (PPG) signals with accelerometer (ACC), gyroscope (GYR), sound, and electrocardiography (ECG) derived smartphone data provides additional insights into the cardiac condition of individuals with and without atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria applicable for all groups:

* At least 18 years old
* Participants must have the ability to understand and provide written informed consent
* Participants must have the ability to understand Dutch

Group specific inclusion criteria:

Group 1: Healthy volunteers

* No cardiac conditions based on medical history.

Group 2: Cardiology patients

* Patients at the consultation or ambulatory unit of Cardiology (pre- cardioversion, pre-pulmonary vein isolation) with AF.
* Patients without AF but with a current cardiac condition (e.g. heart failure with a reduced or preserved ejection fraction) or a history of a cardiac condition (e.g. history of myocardial infarction).

Exclusion Criteria:

* Individuals with unnaturally coloured fingers (i.e. tattoos, ink); this may weaken the signal and may interfere with the effectiveness of the device
* Persons with conditions causing tremors or the inability to hold their hand still for at least 60 seconds (e.g. Parkinson or dementia) as, in this case, the device may not be able to accurately process a measurement
* Persons with reduced blood flow in the fingertips (e.g. perniosis or severe callus formation) as the device may not be able to detect the intensity variations induced by the blood flow
* Persons that have a disability to perform the measurements according to the instructions for use
* Persons with cardiac pacemakers, implantable cardioverter-defibrillators, or other implanted electronic devices as these can control the natural heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of morphologic characteristics of smartphone generated signals | 1 day
  Detect or identify specific morphologic characteristics (changes or correlations) by the comparison of PPG signals, accelerometer signals, gyroscope signals, sound signals and ECG signals, derived via the smartphone data.

SECONDARY OUTCOMES:
Evaluate the performance of the FibriCheck Algorithm | 1 day
  Evaluate the performance of our PPG FibriCheck Algorithm in cardiology patients and healthy volunteers, based on simultaneously recorded ECG data (RR intervals).

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Vandervoort, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium